CLINICAL TRIAL: NCT02109575
Title: Quantitative Detection of Circulating Donor-Specific DNA in Organ Transplant Recipients (DTRT-Multi-Center Study)
Acronym: DTRT
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Columbia University (Other); Duke University (Other); Arkansas Children's Hospital Research Institute (Other); Emory University (Other); Children's Healthcare of Atlanta (Other); Vanderbilt University (Other); TAI Diagnostics, Inc. (Industry); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); University of California, Los Angeles (Other); Children's Hospital Medical Center, Cincinnati (Other); Phoenix Children's Hospital (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Mitchell, Professor Cardiovascular Surgery, Medical College of Wisconsin
Other Study IDs: CHW 10/83; R01HL119747 (NIH)
Record Dates: First submitted 2014-02-10; First posted 2014-04-10 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Disease; Acute Rejection of Cardiac Transplant; Cardiac Transplant Rejection; Heart Transplant Failure and Rejection
Keywords: Acute Rejection; Cardiac Biomarkers; Cardiac Catheterization; Cardiomyopathy; Cell-Free DNA; Congenital Heart Defect; Congenital Heart Disease; Coronary Angiogram; Donor Specific DNA; Donor Specific Cell-Free DNA; Endomyocardial Biopsy; Heart Failure; Heart Transplant Failure; Heart Transplant; Heart Transplant Rejection
MeSH Terms: conditions — Cardiovascular Diseases; Rejection, Psychology; Cardiomyopathies; Heart Defects, Congenital; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Heart Transplant Recipients: Up to 10 cc of blood will be drawn from heart transplant recipients at various time points prior to and after transplant. Blood draw is the only research activity that study participants will undergo. In addition to blood draw, data will be collected from clinical records representing the participant's transplant course such as the medical record, imaging, and biopsy slides with pathology reports.
  Interventions: Diagnostic Test: Blood Draw of up to 10 ml

INTERVENTIONS:
Diagnostic Test: Blood Draw of up to 10 ml — In a laboratory setting, the blood will be spun for plasma and buffy coat, DNA will be extracted for processing using the diagnostic test. The results of the test are not provided back to the clinical setting.

SUMMARY:
The primary goal of this Multicenter Study is to develop and to evaluate a method for measuring donor-specific cell free DNA in blood samples from transplant recipients as markers of rejection. Blood samples obtained periodically from heart transplant recipients are assessed for cell free DNA relative to clinical data in order to determine whether changes in the level of cell free DNA indicate rejection.

This research study proposes testing a blood sample obtained from the heart transplant recipient. The research seeks to establish whether this blood test will show when the patient is beginning to or already rejecting the transplanted heart.

BACKGROUND Identifying if a transplant patient is beginning to or already rejecting the heart is necessary, so that appropriate treatment can be started to halt the rejection. Heart catheterization with biopsy is the usual method used for assessing whether a patient may be rejecting the heart. There are also a number of other methods that transplant physicians will use to look for signs of rejection including other blood tests, echocardiograms, obtaining pressure readings during heart catheterization, and micro-array testing of blood obtained during biopsy. These technologies are limited in ability to consistently and accurately identify the presence of rejection.

The usual method of checking for rejection involves obtaining a sample of the heart tissue (heart biopsy); biopsy can only be accomplished through heart catheterization which is an invasive procedure that has risks associated with disturbing the heart such as puncturing the heart or causing the heart rate to change or damaging tissue in the heart. Overtime, repeating this invasive procedure can diminish the ease of the procedure because the veins can become scarred and more difficult to access. For these reasons, researchers believe that it would be good to have a blood test that gives information about the possibility of rejection so that it may not be necessary to do as many heart biopsies. Also, a blood test may be able to provide information about the heart or about rejection that is currently not available at all.

DETAILED DESCRIPTION:
Early detection of rejection is a major focus of organ transplant care. The use of aggressive immunosuppressive therapy has been shown to alter the prognosis of heart transplant patients who have acute rejection1. There are many modalities utilized in the routine surveillance of heart transplant patients, each with limitations. Screening transthoracic echocardiography focusing on indices of systolic and diastolic dysfunction, along with regional wall abnormalities, has been shown to have poor sensitivity and does not effectively discriminate between patients with and without rejection. Newer echocardiographic parameters including myocardial performance or diastolic velocity indices may be a better means of detecting subtle changes in cardiac function in the setting of heart transplant, but these tools are most helpful after the insult caused by rejection has already occurred. Hemodynamic changes measured during heart catheterization have also been evaluated as a means of detecting rejection. Rosenthal et al found that although there were statistically significant differences between patients with higher or lower grades of rejection scores, heart catheterization did not permit effective discrimination of patients with moderate to severe rejection. Heart biomarkers, including c-reactive protein, brain natriuretic peptides, and troponin, have been studied as non-invasive measures of determining heart dysfunction or rejection. These surrogates are weakly associated with different rejection grades on biopsy and have a poor predictive capacity for biopsy-detected rejection3. Recently, microarray technology has been used to screen for genes expressed in heart allograft rejection using peripheral leukocytes from blood samples obtained at the time of endomyocardial biopsy. This technique was shown to have a high negative predictive value for the diagnosis of acute cellular rejection but it is unable to detect low grades of rejection4. Overall, these technologies are limited in the ability to consistently and accurately predict the presence of rejection and have low positive predictive values when compared to biopsy.

The current gold standard in detection of rejection is the use of endomyocardial biopsy. Attaining these samples is invasive and long term repeated central venous access can be difficult. Risk of endomyocardial biopsy includes perforation leading to cardiac tamponade, arrhythmias including atrial fibrillation, pneumothorax, hemothorax, and valvular regurgitation secondary to rupture of chordae or damage to valve leaflets themselves. There is variability in pathological interpretation of histologic grades, especially at higher grades of rejection due to the difficulty in interpretation of nodular infiltrates. The 2005 revised ISHLT grading system has simplified the grading system of cellular rejection and now includes assessment of antibody mediated rejection. This may improve the utility of endomyocardial biopsy, but much controversy still exists on the method of grading rejection and its clinical implications. Thus, the development of a noninvasive, relatively inexpensive method that accurately predicts the presence of rejection is critical.

ELIGIBILITY:
Inclusion Criteria:

Any patient who is "listed" to undergo or has in the past undergone heart transplantation.

Exclusion Criteria:

Any patient who is not currently listed to undergo heart transplantation or has not previously received a heart transplant;

Any patient who is not anticipated to be available for follow-up of at least 1 year;

Any patient who is unable or unwilling to provide documented informed consent for self or through a legally authorized representative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will include people of any age who have undergone heart transplant or who are "listed" to undergo heart transplant.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Assay and laboratory protocol development and optimization. | Year 1-5
  To develop and optimize an assay and protocol to detect donor-specific cell free DNA from recipient plasma.

SECONDARY OUTCOMES:
Biomarker Development | Year 1-3
  To determine the threshold of elevation of circulating donor specific cell free DNA (cfDNA)

OTHER OUTCOMES:
Validation | Years 4-5
  To validate the threshold and predictive model to evaluate sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mitchell, MD, Principal Investigator — Medical College of Wisconsin; Aoy Tomita-Mitchell, PhD, Principal Investigator — Medical College of Wisconsin
Locations (8):
- United States (8):
  - Arkansas Children's Hosoptial Research Institute, Little Rock, Arkansas
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital Chicago, Chicago, Illinois
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin